CLINICAL TRIAL: NCT05952557
Title: CAMBRIA-2: A Phase III, Open-Label, Randomised Study to Assess the Efficacy and Safety of Camizestrant (AZD9833, a Next Generation, Oral Selective Estrogen Receptor Degrader) vs Standard Endocrine Therapy (Aromatase Inhibitor or Tamoxifen) as Adjuvant Treatment for Patients With ER+/HER2- Early Breast Cancer and an Intermediate-High or High Risk of Recurrence Who Have Completed Definitive Locoregional Treatment and Have No Evidence of Disease
Brief Title: An Adjuvant Endocrine-based Therapy Study of Camizestrant (AZD9833) in ER+/HER2- Early Breast Cancer (CAMBRIA-2)
Acronym: CAMBRIA-2
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Austrian Breast and Colorectal Cancer Study Group (ABCSG) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D8535C00001; 2023-504031-41-00 (Registry Identifier: CTIS (EU))
Record Dates: First submitted 2023-05-17; First posted 2023-07-19 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-06

CONDITIONS: Breast Cancer, Early Breast Cancer
Keywords: ER+; HER2-; breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — AZD9833; Tamoxifen; Anastrozole; Letrozole; exemestane; abemaciclib

STUDY DESIGN:
Intervention Model Description: Patients will be randomised in a 1:1 ratio to one of the following arms: • Arm A: Standard ET of investigator's choice (aromatase inhibitors [AI; exemestane, letrozole, anastrozole] or tamoxifen) ± abemaciclib • Arm B: Camizestrant ± abemaciclib
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A: standard endocrine therapy of investigator´s choice ± abemaciclib (Active Comparator): standard endocrine therapy of investigator's choice (aromatase inhibitors [AI; exemestane, letrozole, anastrozole] or tamoxifen) ± abemaciclib
  Interventions: Drug: Tamoxifen; Drug: Anastrozole; Drug: Letrozole; Drug: Exemestane; Drug: Abemaciclib
- Arm B: camizestrant ± abemaciclib (Experimental): camizestrant ± abemaciclib
  Interventions: Drug: Camizestrant; Drug: Abemaciclib

INTERVENTIONS:
Drug: Camizestrant — Camizestrant. Experimental. Administered orally
  Other Names: AZD9833
  Arms: Arm B: camizestrant ± abemaciclib
Drug: Tamoxifen — Tamoxifen. Comparator. Administered orally
  Arms: Arm A: standard endocrine therapy of investigator´s choice ± abemaciclib
Drug: Anastrozole — Anastrozole. Comparator. Administered orally
  Arms: Arm A: standard endocrine therapy of investigator´s choice ± abemaciclib
Drug: Letrozole — Letrozole. Comparator. Administered orally
  Arms: Arm A: standard endocrine therapy of investigator´s choice ± abemaciclib
Drug: Exemestane — Exemestane. Comparator. Administered orally
  Arms: Arm A: standard endocrine therapy of investigator´s choice ± abemaciclib
Drug: Abemaciclib — Abemaciclib adjuvant treatment Administered orally

SUMMARY:
This is a Phase III open-label study to assess if camizestrant improves outcomes compared to standard adjuvant endocrine therapy for patients with ER+/HER2- early breast cancer with intermediate-high or high risk for disease recurrence who completed definitive locoregional therapy (with or without chemotherapy). The planned duration of treatment in either arm within the study will be 7 years.

DETAILED DESCRIPTION:
This is a Phase III open-label study to assess if camizestrant improves outcomes compared to standard adjuvant endocrine therapy for patients with ER+/HER2- early breast cancer with intermediate-high or high risk for disease recurrence who completed definitive locoregional therapy (with or without chemotherapy). The planned duration of treatment in either arm of the study is 7 years. Eligible patients must have intermediate-high or high risk of recurrence as defined by specified clinical and biologic criteria. Concurrent use of abemaciclib is permitted in both arms. The primary endpoint of the study is Invasive breast cancer-free survival (IBCFS) and main secondary endpoints include Invasive disease-free survival (IDFS), Distant relapse-free survival (DRFS), Overall survival (OS), Safety and Clinical Outcome Assessments (COAs).

Patients will be followed for 10 years from randomization of the last patient.

ELIGIBILITY:
Inclusion Criteria:

* Women and Men; ≥18 years at the time of screening (or per national guidelines)
* Histologically confirmed ER+/HER2- early-stage resected invasive breast cancer with absence of any evidence of metastatic disease as defined in the protocol.
* Completed adequate (definitive) locoregional therapy (surgery with or without radiotherapy) for the primary breast tumour(s), with or without (neo)adjuvant chemotherapy.
* Patients must be randomised within 12 months of definitive breast surgery.
* Patients may have received up to 12 weeks of endocrine therapy prior to randomisation.
* Eastern Cooperative Oncology Group (ECOG) performance status of ≤ 1
* Adequate organ and bone marrow function

Exclusion Criteria:

* Inoperable locally advanced or metastatic breast cancer
* Pathological complete response following treatment with neoadjuvant therapy
* History of any other cancer (except non-melanoma skin cancer or carcinoma in situ of the cervix or considered a very low risk of recurrence per investigator judgement) unless in complete remission with no therapy for a minimum of 5 years from the date of randomisation
* Any evidence of severe or uncontrolled systemic diseases which, in the investigator's opinion precludes participation in the study or compliance "
* Known LVEF <50% with heart failure NYHA Grade ≥2.
* Mean resting QTcF interval > 480 ms at screening
* Concurrent exogenous reproductive hormone therapy or non topical hormonal therapy for non-cancer-related conditions
* Any concurrent anti-cancer treatment not specified in the protocol with the exception of bisphosphonates (e.g. zoledronic acid) or RANKL inhibitors ( eg, denosumab)
* Previous treatment with camizestrant, investigational SERDs/investigational ER targeting agents, or fulvestrant
* Currently pregnant (confirmed with positive serum pregnancy test) or breastfeeding.
* Patients with known hypersensitivity to active or inactive excipients of camizestrant or drugs with a similar chemical structure or class to camizestrant. In pre-/peri-menopausal female and male patients, known hypersensitivity or intolerance to LHRH agonists that would preclude the patient from receiving any LHRH agonist.

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5500 (Estimated)
Dates: Start 2023-10-05 (Actual); Primary Completion 2030-03-04 (Estimated); Study Completion 2037-05-06 (Estimated)

PRIMARY OUTCOMES:
Invasive breast cancer-free survival (IBCFS) | Up to 14 years
  IBCFS is defined as time from randomisation until date of first occurrence of:
  * Invasive ipsilateral breast tumour recurrence
  * Locoregional invasive breast cancer recurrence
  * Distant recurrence
  * Contralateral invasive breast cancer
  * Death attributable to any cause.

SECONDARY OUTCOMES:
Invasive disease-free survival (IDFS) | Up to 14 years
  IDFS is defined as time from randomisation until date of first occurrence of one of the following events:
  * Invasive ipsilateral breast tumor recurrence
  * Locoregional invasive breast cancer recurrence
  * Distant recurrence
  * Contralateral invasive breast cancer
  * Second primary non-breast invasive cancer
  * Death attributable to any cause.
Distant relapse-free survival (DRFS) | Up to 14 years
  DRFS is defined as time from randomisation until date of first distant recurrence or death from any cause, whichever occurs first.
Overall survival (OS) | Up to 14 years
  OS is defined as time from randomisation until death from any cause.
Incidence and Severity of Adverse Events, with Severity Determined According to National Cancer Institute Common Terminology Criteria for Adverse Events, version 5.0 (NCI-CTCAE v5.0) | Until 28 days after the final dose of study treatment (up to 7 years)
Proportion of time on study treatment with high side-effect burden as measured by the PGI-TT. | Until 28 days after the final dose of study treatment (up to 7 years)
Change from baseline and time to deterioration of health-related quality of life as measured by the 2 global QoL items from the EORTC IL-311 | Until 28 days after the final dose of study treatment (up to 7 years)
Pharmacokinetics (PK) | Until 6 months from treatment start
  Plasma concentrations of camizestrant pre-dose (trough concentration)

CONTACTS AND LOCATIONS:
Locations (634):
- United States (131):
  - Research Site, Dothan, Alabama
  - Research Site, Phoenix, Arizona
  - Research Site, Tucson, Arizona
  - Research Site, Fayetteville, Arkansas
  - Research Site, Duarte, California
  - Research Site, Fountain Valley, California
  - Research Site, Greenbrae, California
  - Research Site, Irvine, California
  - Research Site, La Jolla, California
  - Research Site, Los Angeles, California
  - Research Site, Monterey, California
  - Research Site, Walnut Creek, California
  - Research Site, West Hollywood, California
  - Research Site, Aurora, Colorado
  - Research Site, Littleton, Colorado
  - Research Site, New Haven, Connecticut
  - Research Site, Newark, Delaware
  - Research Site, Washington D.C., District of Columbia
  - Research Site, Clearwater, Florida
  - Research Site, Fort Myers, Florida
  - Research Site, Gainesville, Florida
  - Research Site, Jacksonville, Florida
  - Research Site, Orlando, Florida
  - Research Site, Pembroke Pines, Florida
  - Research Site, Plantation, Florida
  - Research Site, St. Petersburg, Florida
  - Research Site, Tallahassee, Florida
  - Research Site, West Palm Beach, Florida
  - Research Site, Atlanta, Georgia
  - Research Site, Columbus, Georgia
  - Research Site, Marietta, Georgia
  - Research Site, Savannah, Georgia
  - Research Site, Thomasville, Georgia
  - Research Site, Chicago, Illinois
  - Research Site, Elmhurst, Illinois
  - Research Site, Naperville, Illinois
  - Research Site, Park Ridge, Illinois
  - Research Site, Plainfield, Illinois
  - Research Site, Urbana, Illinois
  - Research Site, Fort Wayne, Indiana
  - Research Site, Des Moines, Iowa
  - Research Site, Fairway, Kansas
  - Research Site, Louisville, Kentucky
  - Research Site, New Orleans, Louisiana
  - Research Site, Scarborough, Maine
  - Research Site, Annapolis, Maryland
  - Research Site, Baltimore, Maryland
  - Research Site, Bethesda, Maryland
  - Research Site, Lutherville, Maryland
  - Research Site, Towson, Maryland
  - Research Site, Boston, Massachusetts
  - Research Site, Hyannis, Massachusetts
  - Research Site, Worcester, Massachusetts
  - Research Site, Detroit, Michigan
  - Research Site, Flint, Michigan
  - Research Site, Ypsilanti, Michigan
  - Research Site, Minneapolis, Minnesota
  - Research Site, Rochester, Minnesota
  - Research Site, Kansas City, Missouri
  - Research Site, St Louis, Missouri
  - Research Site, Lincoln, Nebraska
  - Research Site, Omaha, Nebraska
  - Research Site, Hooksett, New Hampshire
  - Research Site, Lebanon, New Hampshire
  - Research Site, Manchester, New Hampshire
  - Research Site, New Brunswick, New Jersey
  - Research Site, Albuquerque, New Mexico
  - Research Site, Farmington, New Mexico
  - Research Site, Bay Shore, New York
  - Research Site, East Syracuse, New York
  - Research Site, Greenlawn, New York
  - Research Site, New Hyde Park, New York
  - Research Site, New York, New York
  - Research Site, Stony Brook, New York
  - Research Site, White Plains, New York
  - Research Site, Charlotte, North Carolina
  - Research Site, Durham, North Carolina
  - Research Site, Greensboro, North Carolina
  - Research Site, Greenville, North Carolina
  - Research Site, Pinehurst, North Carolina
  - Research Site, Raleigh, North Carolina
  - Research Site, Winston-Salem, North Carolina
  - Research Site, Blue Ash, Ohio
  - Research Site, Cincinnati, Ohio
  - Research Site, Cleveland, Ohio
  - Research Site, Columbus, Ohio
  - Research Site, Toledo, Ohio
  - Research Site, Youngstown, Ohio
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, Portland, Oregon
  - Research Site, Gettysburg, Pennsylvania
  - Research Site, Hershey, Pennsylvania
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Pittsburgh, Pennsylvania
  - Research Site, Sayre, Pennsylvania
  - Research Site, York, Pennsylvania
  - Research Site, Charleston, South Carolina
  - Research Site, Greenville, South Carolina
  - Research Site, Rock Hill, South Carolina
  - Research Site, Spartanburg, South Carolina
  - Research Site, Aberdeen, South Dakota
  - Research Site, Sioux Falls, South Dakota
  - Research Site, Chattanooga, Tennessee
  - Research Site, Knoxville, Tennessee
  - Research Site, Memphis, Tennessee
  - Research Site, Nashville, Tennessee
  - Research Site, Austin, Texas
  - Research Site, Bedford, Texas
  - Research Site, Dallas, Texas
  - Research Site, El Paso, Texas
  - Research Site, Flower Mound, Texas
  - Research Site, Houston, Texas
  - Research Site, Plano, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Tyler, Texas
  - Research Site, Salt Lake City, Utah
  - Research Site, Charlottesville, Virginia
  - Research Site, Fairfax, Virginia
  - Research Site, Midlothian, Virginia
  - Research Site, Norfolk, Virginia
  - Research Site, Richmond, Virginia
  - Research Site, Roanoke, Virginia
  - Research Site, Winchester, Virginia
  - Research Site, Puyallup, Washington
  - Research Site, Spokane, Washington
  - Research Site, Vancouver, Washington
  - Research Site, Charleston, West Virginia
  - Research Site, Morgantown, West Virginia
  - Research Site, Appleton, Wisconsin
  - Research Site, Madison, Wisconsin
  - Research Site, Milwaukee, Wisconsin
- Argentina (9):
  - Research Site, Buenos Aires
  - Research Site, CABA
  - Research Site, Capital Federal
  - Research Site, Córdoba
  - Research Site, La Plata
  - Research Site, Rosario
  - Research Site, San Juan
  - Research Site, San Miguel de Tucumán
  - Research Site, Viedma
- Australia (26):
  - Research Site, Adelaide
  - Research Site, Bankstown
  - Research Site, Bendigo
  - Research Site, Bowral
  - Research Site, Brighton
  - Research Site, Clayton
  - Research Site, Coffs Harbour
  - Research Site, Fitzroy
  - Research Site, Frankston
  - Research Site, Garran
  - Research Site, Gateshead
  - Research Site, Heidelberg
  - Research Site, Liverpool
  - Research Site, Melbourne
  - Research Site, Murdoch
  - Research Site, Randwick
  - Research Site, Richmond
  - Research Site, Shepparton
  - Research Site, South Brisbane
  - Research Site, St Leonards
  - Research Site, Subiaco
  - Research Site, Traralgon
  - Research Site, Wangaratta
  - Research Site, Waratah
  - Research Site, Warnnambool
  - Research Site, Wollongong
- Austria (10):
  - Research Site, Graz
  - Research Site, Innsbruck
  - Research Site, Klagenfurt
  - Research Site, Linz
  - Research Site, Salzburg
  - Research Site, Sankt Veit an der Glan
  - Research Site, Steyr
  - Research Site, Vienna
  - Research Site, Wels
  - Research Site, Wiener Neustadt
- Belgium (10):
  - Research Site, Aalst
  - Research Site, Anderlecht
  - Research Site, Brasschaat
  - Research Site, Brussels
  - Research Site, Charleroi
  - Research Site, Edegem
  - Research Site, Ghent
  - Research Site, Leuven
  - Research Site, Namur
  - Research Site, Wilrijk
- Brazil (23):
  - Research Site, Alfenas
  - Research Site, Belo Horizonte
  - Research Site, Blumenau
  - Research Site, Brasília
  - Research Site, Curitiba
  - Research Site, Fortaleza
  - Research Site, Goiânia
  - Research Site, Itajaí
  - Research Site, João Pessoa
  - Research Site, Natal
  - Research Site, Porto Alegre
  - Research Site, Porto Velho
  - Research Site, Pouso Alegre
  - Research Site, Recife
  - Research Site, Ribeirão Preto
  - Research Site, Rio de Janeiro
  - Research Site, Salvador
  - Research Site, Santo André
  - Research Site, São Paulo
  - Research Site, Taubaté
  - Research Site, Teresina
  - Research Site, Três Lagoas
  - Research Site, Vitória
- Bulgaria (7):
  - Research Site, Dobrich
  - Research Site, Haskovo
  - Research Site, Plovdiv
  - Research Site, Shumen
  - Research Site, Sofia
  - Research Site, Varna
  - Research Site, Vratsa
- Canada (16):
  - Research Site, Calgary, Alberta
  - Research Site, Edmonton, Alberta
  - Research Site, Kelowna, British Columbia
  - Research Site, North Vancouver, British Columbia
  - Research Site, Halifax, Nova Scotia
  - Research Site, Barrie, Ontario
  - Research Site, Greater Sudbury, Ontario
  - Research Site, Kingston, Ontario
  - Research Site, Sault Ste. Marie, Ontario
  - Research Site, Thunder Bay, Ontario
  - Research Site, Windsor, Ontario
  - Research Site, Chicoutimi, Quebec
  - Research Site, Lévis, Quebec
  - Research Site, Montreal, Quebec
  - Research Site, Québec, Quebec
  - Research Site, Saskatoon, Saskatchewan
- Chile (7):
  - Research Site, Concepción
  - Research Site, La Serena
  - Research Site, Port Montt
  - Research Site, Providencia
  - Research Site, Santiago
  - Research Site, Temuco
  - Research Site, Viña del Mar
- China (46):
  - Research Site, Baoding
  - Research Site, Beijing
  - Research Site, Bengbu
  - Research Site, Binzhou
  - Research Site, Cangzhou
  - Research Site, Changchun
  - Research Site, Changsha
  - Research Site, Chengdu
  - Research Site, Chifeng
  - Research Site, Dalian
  - Research Site, Foshan
  - Research Site, Fuzhou
  - Research Site, Guangzhou
  - Research Site, Haikou
  - Research Site, Hangzhou
  - Research Site, Harbin
  - Research Site, Hefei
  - Research Site, Hohhot
  - Research Site, Huizhou
  - Research Site, Jinzhou
  - Research Site, Lanzhou
  - Research Site, Linyi
  - Research Site, Liuchow
  - Research Site, Nanchang
  - Research Site, Nanjing
  - Research Site, Nanning
  - Research Site, Nantong
  - Research Site, Neijiang
  - Research Site, Shandong
  - Research Site, Shangqiu
  - Research Site, Shantou
  - Research Site, Shaoguan Shi
  - Research Site, Shenyang
  - Research Site, Shenzhen
  - Research Site, Shijiazhuang
  - Research Site, Suining Shi
  - Research Site, Suzhou
  - Research Site, Taizhou
  - Research Site, Tianjin
  - Research Site, Weifang
  - Research Site, Wuhan
  - Research Site, Xi'an
  - Research Site, Xiangfan
  - Research Site, Xinxiang
  - Research Site, Xuzhou
  - Research Site, Zunyi
- Colombia (6):
  - Research Site, Barranquilla
  - Research Site, Bogotá
  - Research Site, Cali
  - Research Site, Medellín
  - Research Site, Montería
  - Research Site, Valledupar
- Croatia (5):
  - Research Site, Osijek
  - Research Site, Rijeka
  - Research Site, Split
  - Research Site, Zadar
  - Research Site, Zagreb
- Czechia (5):
  - Research Site, Brno
  - Research Site, Hořovice
  - Research Site, Liberec
  - Research Site, Pardubice
  - Research Site, Prague
- Estonia (2):
  - Research Site, Tallinn
  - Research Site, Tartu
- France (24):
  - Research Site, Angers
  - Research Site, Bordeaux
  - Research Site, Caen
  - Research Site, Clermont-Ferrand
  - Research Site, Dijon
  - Research Site, Epagny Metz-Tessy
  - Research Site, Lille
  - Research Site, Lyon
  - Research Site, Marseille
  - Research Site, Montpellier
  - Research Site, Nantes
  - Research Site, Nîmes
  - Research Site, Paris
  - Research Site, Pierre-Bénite
  - Research Site, Plerin SUR MER
  - Research Site, Rennes
  - Research Site, Rouen
  - Research Site, Saint-Cloud
  - Research Site, Saint-Herblain
  - Research Site, Saint-Priest-en-Jarez
  - Research Site, Strasbourg
  - Research Site, Toulouse
  - Research Site, Vandœuvre-lès-Nancy
  - Research Site, Villejuif
- Georgia (2):
  - Research Site, Batumi
  - Research Site, Tbilisi
- Germany (30):
  - Research Site, Aachen
  - Research Site, Berlin
  - Research Site, Cologne
  - Research Site, Darmstadt
  - Research Site, Deggendorf
  - Research Site, Dessau
  - Research Site, Dresden
  - Research Site, Düsseldorf
  - Research Site, Essen
  - Research Site, Freudenstadt
  - Research Site, Georgsmarienhütte
  - Research Site, Hamburg
  - Research Site, Hamm
  - Research Site, Hanau
  - Research Site, Hanover
  - Research Site, Heidelberg
  - Research Site, Karlsruhe
  - Research Site, Koblenz
  - Research Site, Mainz
  - Research Site, Nürtingen
  - Research Site, Offenburg
  - Research Site, Rostock
  - Research Site, Saarbrücken
  - Research Site, Schweinfurt
  - Research Site, Speyer
  - Research Site, Torgau
  - Research Site, Wiesbaden
  - Research Site, Witten
  - Research Site, Worms
  - Research Site, Wuppertal
- Greece (8):
  - Research Site, Athens
  - Research Site, Heraklion
  - Research Site, Ioannina
  - Research Site, Larissa
  - Research Site, Marousi
  - Research Site, Piraeus
  - Research Site, Rio
  - Research Site, Thessaloniki
- Hungary (12):
  - Research Site, Budapest
  - Research Site, Debrecen
  - Research Site, Győr
  - Research Site, Gyula
  - Research Site, Kaposvár
  - Research Site, Kecskemét
  - Research Site, Miskolc
  - Research Site, Nyíregyháza
  - Research Site, Salgótarján
  - Research Site, Szeged
  - Research Site, Szekszárd
  - Research Site, Zalaegerszeg
- India (18):
  - Research Site, Ansārinagar
  - Research Site, Bangalore
  - Research Site, Belgavi
  - Research Site, Dehradun
  - Research Site, Delhi
  - Research Site, Dhanvantari Nagar
  - Research Site, Gūrgaon
  - Research Site, Hyderabad
  - Research Site, Jaipur
  - Research Site, Kanpur
  - Research Site, Kolkata
  - Research Site, Kozhikode
  - Research Site, Mumbai
  - Research Site, Mysuru
  - Research Site, Nagpur
  - Research Site, Nashik
  - Research Site, New Delhi
  - Research Site, Surat
- Ireland (4):
  - Research Site, Cork
  - Research Site, Dublin
  - Research Site, Galway
  - Research Site, Waterford
- Israel (8):
  - Research Site, Afula
  - Research Site, Ashdod
  - Research Site, Beersheba
  - Research Site, Haifa
  - Research Site, Jerusalem
  - Research Site, Kfar Saba
  - Research Site, Nahariya
  - Research Site, Ramat Gan
- Italy (17):
  - Research Site, Bergamo
  - Research Site, Bologna
  - Research Site, Brindisi
  - Research Site, Florence
  - Research Site, Genoa
  - Research Site, Meldola
  - Research Site, Milan
  - Research Site, Misterbianco
  - Research Site, Modena
  - Research Site, Monza
  - Research Site, Napoli
  - Research Site, Novara
  - Research Site, Padua
  - Research Site, Roma
  - Research Site, Rozzano
  - Research Site, Torino
  - Research Site, Trento
- Japan (28):
  - Research Site, Bunkyō City
  - Research Site, Chiba
  - Research Site, Chūōku
  - Research Site, Fukuoka
  - Research Site, Fukushima
  - Research Site, Hirakata-shi
  - Research Site, Hiroshima
  - Research Site, Iruma-Gun
  - Research Site, Isehara-shi
  - Research Site, Kagoshima
  - Research Site, Kashiwa
  - Research Site, Kōtoku
  - Research Site, Kumamoto
  - Research Site, Kurume-shi
  - Research Site, Kyoto
  - Research Site, Matsuyama
  - Research Site, Nagoya
  - Research Site, Niigata
  - Research Site, Osaka
  - Research Site, Ota-shi
  - Research Site, Sapporo
  - Research Site, Sendai
  - Research Site, Shinagawa-ku
  - Research Site, Suita-shi
  - Research Site, Sunto-gun
  - Research Site, Takasaki-shi
  - Research Site, Tsu
  - Research Site, Yokohama
- Malaysia (6):
  - Research Site, Johor Bahru
  - Research Site, Kota Bharu
  - Research Site, Kuala Lumpur
  - Research Site, Kuching
  - Research Site, Malacca
  - Research Site, Pulau Pinang
- Mexico (10):
  - Research Site, Alc. Cuauhtémoc
  - Research Site, Cancún
  - Research Site, Colonia Lindavista
  - Research Site, Estado de México
  - Research Site, Mérida
  - Research Site, México
  - Research Site, Monterrey
  - Research Site, San Luis Potosí City
  - Research Site, Tuxtla Gutiérrez
  - Research Site, Veracruz
- New Zealand (3):
  - Research Site, Auckland
  - Research Site, Hamilton
  - Research Site, Palmerston North
- Peru (5):
  - Research Site, Arequipa
  - Research Site, La Libertad
  - Research Site, Lima
  - Research Site, San Isidro
  - Research Site, Trujillo
- Philippines (5):
  - Research Site, Bacolod
  - Research Site, Cebu City
  - Research Site, Iloilo City
  - Research Site, Manila
  - Research Site, Quezon
- Poland (18):
  - Research Site, Bialystok
  - Research Site, Biała Podlaska
  - Research Site, Bydgoszcz
  - Research Site, Gdansk
  - Research Site, Gdynia
  - Research Site, Grudziądz
  - Research Site, Koszalin
  - Research Site, Krakow
  - Research Site, Lodz
  - Research Site, Lublin
  - Research Site, Opole
  - Research Site, Poznan
  - Research Site, Racibórz
  - Research Site, Rzeszów
  - Research Site, Szczecin
  - Research Site, Tomaszów Mazowiecki
  - Research Site, Warsaw
  - Research Site, Wroclaw
- Portugal (8):
  - Research Site, Amadora
  - Research Site, Braga
  - Research Site, Lisbon
  - Research Site, Matosinhos Municipality
  - Research Site, Porto
  - Research Site, Viana do Castelo
  - Research Site, Vila Nova de Gaia
  - Research Site, Vila Real
- Research Site, Rio Piedras, Puerto Rico
- Romania (11):
  - Research Site, Bucharest
  - Research Site, Cluj-Napoca
  - Research Site, Craiova
  - Research Site, Floreşti
  - Research Site, Iași
  - Research Site, Oradea
  - Research Site, Otopeni
  - Research Site, Ovidiu
  - Research Site, Piteşti
  - Research Site, Sibiu
  - Research Site, Timișoara
- Saudi Arabia (2):
  - Research Site, Riyadh
  - Research Site, Riyadh/MENA
- Serbia (6):
  - Research Site, Belgrade
  - Research Site, Kragujevac
  - Research Site, Niš
  - Research Site, Novi Sad
  - Research Site, Valjevo
  - Research Site, Zrenjanin
- South Africa (8):
  - Research Site, Bloemfontein
  - Research Site, Cape Town
  - Research Site, eManzimtoti
  - Research Site, George
  - Research Site, Johannesburg
  - Research Site, Pietermaritzburg
  - Research Site, Port Elizabeth
  - Research Site, Pretoria
- South Korea (5):
  - Research Site, Cheonan-si
  - Research Site, Daegu
  - Research Site, Goyang-si
  - Research Site, Seongnam-si
  - Research Site, Seoul
- Spain (34):
  - Research Site, A Coruña
  - Research Site, Albacete
  - Research Site, Alicante
  - Research Site, Badalona
  - Research Site, Barakaldo
  - Research Site, Barcelona
  - Research Site, Burgos
  - Research Site, Castellon
  - Research Site, Cáceres
  - Research Site, Córdoba
  - Research Site, Donostia / San Sebastian
  - Research Site, El Palmar
  - Research Site, Elche(Alicante)
  - Research Site, Fuenlabrada
  - Research Site, Girona
  - Research Site, Granada
  - Research Site, Jerez de la Frontera
  - Research Site, La Laguna (Tenerife)
  - Research Site, León
  - Research Site, Lleida
  - Research Site, Madrid
  - Research Site, Manresa
  - Research Site, Málaga
  - Research Site, Murcia
  - Research Site, Palma de Mallorca
  - Research Site, Reus,Tarragona
  - Research Site, Sabadell
  - Research Site, Salamanca
  - Research Site, Sant Joan Despí
  - Research Site, Seville
  - Research Site, Toledo
  - Research Site, Valencia
  - Research Site, Vigo
  - Research Site, Zaragoza
- Switzerland (11):
  - Research Site, Baden
  - Research Site, Basel
  - Research Site, Bellinzona
  - Research Site, Chur
  - Research Site, Frauenfeld
  - Research Site, La Chaux-de-Fonds
  - Research Site, Lausanne
  - Research Site, Lucerne
  - Research Site, Sankt Gallen
  - Research Site, Winterthur
  - Research Site, Zurich
- Taiwan (7):
  - Research Site, Hsinchu
  - Research Site, Kaohsiung City
  - Research Site, New Taipei City
  - Research Site, Taichung
  - Research Site, Tainan
  - Research Site, Taipei
  - Research Site, Yongkang District
- Thailand (3):
  - Research Site, Bangkok
  - Research Site, Hat Yai
  - Research Site, Khon Kaen
- Turkey (Türkiye) (10):
  - Research Site, Ankara
  - Research Site, Antalya
  - Research Site, Bursa
  - Research Site, Çankaya
  - Research Site, Çiğli
  - Research Site, Edirne
  - Research Site, Istanbul
  - Research Site, Karşıyaka
  - Research Site, Malatya
  - Research Site, Samsun
- United Arab Emirates (3):
  - Research Site, Abu Dhabi
  - Research Site, Al Ain City
  - Research Site, Dubai
- United Kingdom (24):
  - Research Site, Aberdeen
  - Research Site, Bath
  - Research Site, Brighton
  - Research Site, Burton-on-Trent
  - Research Site, Cambridge
  - Research Site, Derby
  - Research Site, Guildford
  - Research Site, Ipswich
  - Research Site, Lancaster
  - Research Site, Leeds
  - Research Site, Leicester
  - Research Site, Liverpool
  - Research Site, London
  - Research Site, Manchester
  - Research Site, Northampton
  - Research Site, Oxford
  - Research Site, Reading
  - Research Site, Shrewsbury
  - Research Site, Stockton
  - Research Site, Sutton
  - Research Site, Sutton in Ashfield
  - Research Site, Taunton
  - Research Site, Warwick
  - Research Site, Whitchurch

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please refer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool. Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Derived] Hamilton EP, Loibl S, Bachelot T, Gnant M, Niikura N, Park YH, Tolaney SM, Pistilli B, Rastogi P, Saini KS, Gioni I, Johnston S, Nunes R, Quintana A, Stuart M, Syta E, Walding A, Klinowska T, Mayer IA. CAMBRIA-1 & CAMBRIA-2 phase III trials: camizestrant versus standard endocrine therapy in ER+/HER2- early breast cancer. Future Oncol. 2025 Mar;21(7):795-806. doi: 10.1080/14796694.2025.2459548. Epub 2025 Feb 27. PMID 40017004
- See also: Breast Cancer Study Locator details (for US) — https://www.breastcancerstudylocator.com/trial/listing/411695